CLINICAL TRIAL: NCT02472899
Title: Peripheral Markers of Inflammation in Patients With Alzheimer's Disease Compared to Cognitively Normal Elderly
Brief Title: Biomarker Study for Alzheimer's Disease
Acronym: BiomarkerAD
Status: Completed | Type: Observational
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Principal Investigator, Beersheva Mental Health Center
Other Study IDs: CT4525
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer's Disease
Keywords: Geriatrics; Neurocognitive Disorder; Biomarkers; Immunology
MeSH Terms: conditions — Alzheimer Disease; Neurocognitive Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Frozen serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alzheimer's Disease: Blood sample from subjects older than 60 years with a clinical diagnosis of Alzheimer's Disease
  Interventions: Other: Blood sample
- Older controls: Blood sample from subjects older than 60 years who are cognitively normal
  Interventions: Other: Blood sample
- Younger controls: Blood sample from healthy subjects aged 20 to 30 years who are cognitively normal
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Non-interventional study based on blood samples taken at a single study visit

SUMMARY:
The study aims to identify immune biomarkers in peripheral blood for identifying Alzheimer's disease (AD). Blood samples from subjects with AD will be compared to age-matched controls without cognitive symptoms, as well as healthy younger subjects.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive neurodegenerative disease characterized by the loss of cognitive brain functions and functional decline. One of the pathological features of this condition is the progressive deposition in the brain of amyloid beta-peptide (A-beta) (1). Once deposited in the brain, the peptide exerts a toxic effect by triggering a chronic inflammation that interferes initially with normal brain function and results eventually in neuronal death (2). It is currently postulated that at a certain threshold of A-beta accumulation compensatory mechanisms in the brain are no longer sufficient to cope with A-beta toxicity, and the clinical syndrome of AD develops. It is possible that A-beta may accumulate in the brain over a period of up to 10-15 years before clinical symptoms become significant. The question has been raised whether the accumulation of A-beta is possibly a normal process of aging, suggesting that all people may be susceptible to the disease if they live long enough - of note is that the prevalence of Alzheimer's disease rises to over 40% above the age of 85 years.

Among the many possible ageing-related factors involved in the development of AD, senescence of the immune system may significantly enhance changes in the brain and intensify the neurological decline in patients with this disease. A direct consequence of immunosenescence is the increased frequency of systemic infections and, in fact, many who die with AD have previously suffered from a severe infection. Since patients with AD have an ongoing chronic inflammatory response in the brain, associated with the activation of glial cells and a partially disrupted blood brain barrier, systemic inflammation may intensify this process in the brain and increase the overall neuronal damage.

In contrast to the damage caused by immune activation, A-beta vaccination studies have shown very promising effects in mouse models of the disease, particularly with regard to the clearance of amyloid plaques by A-beta antibodies (3). When tested in patients with AD, 6% of the vaccinated patients developed severe inflammatory reactions in the brain (4). Nonetheless, a cohort of patients showed improved cognitive tests where specific antibodies were induced (5). In a recent study we demonstrated that such brain inflammation may be due to increased levels of IFN-γ in the brain (6), possibly as a result of sub-clinical systemic infection and the specific immune responses observed in humans.

While the chronic inflammation progresses throughout the disease, the specific arm of the immune system, i.e., brain-specific lymphocytes, may also be stimulated to play a role. In contrast to previous assumptions, our findings in human subjects with AD demonstrate that a specific immune response to A-beta is indeed significantly induced in both elderly individuals and patients with AD as compared to middle-aged individuals (7). The nature and role of this immune response to A-beta in man is yet to be investigated, and may lead to the characterization of pathways associated with neuronal cell death, and result in new diagnostic modalities and immunotherapeutic approaches.

The purpose of this study is to determine whether peripheral markers possibly related to A-beta induced inflammation of the brain are increased in patients with clinical AD.

Method This is an observational pilot study comparing the level of inflammatory markers in the peripheral blood of patients with AD to that of age-matched and cognitively normal elderly individuals, as well as to healthy young controls.

Subjects will include males and females older than 60 years diagnosed as having clinical AD according to DSM-IV criteria. The control group will comprise cognitively normal community dwelling males and females older than 60 years. In addition, a group of healthy young male and female controls aged 20-30 years will serve as the reference group. The diagnosis of both older patients and controls will be determined independently by a multidisciplinary team of experts at the Memory Clinic of the Beersheva Mental Health Center.

All subjects and controls will be required to provide written informed consent for participation in the study. In the case of the patients with AD an independent psychiatrist will be required to confirm that the patient is capable of agreeing to participation in the study. In the case of patients with AD who have impaired judgment and are unable to consent to their participation, a legal guardian will be required to provide written informed consent.

Following the acquisition of demographic data, a single amount of 25 ml of blood will be drawn from all subjects. Blood will be drawn into two heparinized tubes of 10 ml each and one serological tube (with procoagulant) of five ml will be drawn for serum isolation. The heparinized tubes will be maintained at room temperature until lymphocytes are purified on the same day. Sera samples will be stored at 4°C. Blood will be drawn before midday to facilitate purification on the same day. Following peripheral blood mononuclear cell (PBMC) and sera isolation the following analysis will be performed:

1. Generation of AD-specific monoclonal antibodies. Since antibodies which bind the N-terminus portion of A-beta enhance its clearance from the brain and are now tested in a clinical trial, it is important to identify the naturally occurring specific monoclonal antibodies induced in patients with AD and determine whether they affect the course of the disease. Such specific antibodies also may have diagnostic and therapeutic properties. These specific human monoclonal antibodies will be isolated and produced in vitro by the hybridoma technique using a proprietary fusion partner cell line known as MFP-2. Briefly, PBMCs will be fused with MFP-2 and the resulting hybridomas will be screened for nonspecific Ig production and then for those immunoglobulins that are specific to A-beta using standard techniques of ELISA. Hybridomas that secrete specific human monoclonal antibodies will be serially subcloned for stabilization, expanded and grown in defined media for production of large quantities of monoclonal antibodies.
2. Analysis of T-cell subsets and serum-derived cytokines. Aging is associated with senecense of the immune system expressed by a decline in naïve T cells and an increase in memory and regulatory T cells. As a result cytokine homeostasis both in the periphery and in the brain is altered and may contribute to the pathogenesis of AD. Thus, analysis of T-cell subsets (naïve and memory CD4, CD8, and regulatory CD4CD25) using Fluorescence-activated cell sorting (FACS) and serum-derived cytokines by ELISA will be performed and correlated with the clinical score of the patients.

Statistical evaluation of differences in mean values between groups will be performed using the Student's-t test.

ELIGIBILITY:
Inclusion Criteria:

* Dementia syndrome resulting from probable Alzheimer's disease

Exclusion Criteria:

* Dementia syndrome caused by conditions other than Alzheimer's disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will include males and females older than 60 years diagnosed as having clinical AD according to DSM-IV criteria. The control group will comprise cognitively normal community dwelling males and females older than 60 years. In addition, a group of healthy young male and female controls aged 20-30 years will serve as the reference group. The diagnosis of both older patients and controls will be determined independently by a multidisciplinary team of experts at the Memory Clinic of the Beersheva Mental Health Center.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2007-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Frequency of monoclonal antibodies and of CD4+ and CD25+ T cells | Up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD, Principal Investigator — Beersheva Mental Health Center
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel

REFERENCES:
- [Background] Selkoe DJ. Alzheimer's disease: genes, proteins, and therapy. Physiol Rev. 2001 Apr;81(2):741-66. doi: 10.1152/physrev.2001.81.2.741. PMID 11274343
- [Background] McGeer PL, Rogers J, McGeer EG. Inflammation, anti-inflammatory agents and Alzheimer disease: the last 12 years. J Alzheimers Dis. 2006;9(3 Suppl):271-6. doi: 10.3233/jad-2006-9s330. PMID 16914866
- [Background] Schenk D, Barbour R, Dunn W, Gordon G, Grajeda H, Guido T, Hu K, Huang J, Johnson-Wood K, Khan K, Kholodenko D, Lee M, Liao Z, Lieberburg I, Motter R, Mutter L, Soriano F, Shopp G, Vasquez N, Vandevert C, Walker S, Wogulis M, Yednock T, Games D, Seubert P. Immunization with amyloid-beta attenuates Alzheimer-disease-like pathology in the PDAPP mouse. Nature. 1999 Jul 8;400(6740):173-7. doi: 10.1038/22124. PMID 10408445
- [Background] Orgogozo JM, Gilman S, Dartigues JF, Laurent B, Puel M, Kirby LC, Jouanny P, Dubois B, Eisner L, Flitman S, Michel BF, Boada M, Frank A, Hock C. Subacute meningoencephalitis in a subset of patients with AD after Abeta42 immunization. Neurology. 2003 Jul 8;61(1):46-54. doi: 10.1212/01.wnl.0000073623.84147.a8. PMID 12847155
- [Background] Hock C, Konietzko U, Streffer JR, Tracy J, Signorell A, Muller-Tillmanns B, Lemke U, Henke K, Moritz E, Garcia E, Wollmer MA, Umbricht D, de Quervain DJ, Hofmann M, Maddalena A, Papassotiropoulos A, Nitsch RM. Antibodies against beta-amyloid slow cognitive decline in Alzheimer's disease. Neuron. 2003 May 22;38(4):547-54. doi: 10.1016/s0896-6273(03)00294-0. PMID 12765607
- [Background] Monsonego A, Imitola J, Petrovic S, Zota V, Nemirovsky A, Baron R, Fisher Y, Owens T, Weiner HL. Abeta-induced meningoencephalitis is IFN-gamma-dependent and is associated with T cell-dependent clearance of Abeta in a mouse model of Alzheimer's disease. Proc Natl Acad Sci U S A. 2006 Mar 28;103(13):5048-53. doi: 10.1073/pnas.0506209103. Epub 2006 Mar 20. PMID 16549802
- [Background] Monsonego A, Zota V, Karni A, Krieger JI, Bar-Or A, Bitan G, Budson AE, Sperling R, Selkoe DJ, Weiner HL. Increased T cell reactivity to amyloid beta protein in older humans and patients with Alzheimer disease. J Clin Invest. 2003 Aug;112(3):415-22. doi: 10.1172/JCI18104. PMID 12897209